# PARTNERS HUMAN RESEARCH COMMITTEE DETAILED PROTOCOL

Electronic Tools to Increase Recognition and Improve Primary Care Management for Hypertension in Chronic Kidney Disease

P.I.: Lipika Samal M.D., M.P.H.

#### I. BACKGROUND AND SIGNIFIGANCE

Prevalence, Outcomes and Cost of Chronic Kidney Disease: Chronic kidney disease (CKD) is prevalent, afflicting 26 million Americans, and is a condition associated with high morbidity and mortality. In addition, CKD is costly. The average cost per person per year is about \$20,000 and Medicare costs for ESRD total \$26.8 billion. CKD Diagnosis, Monitoring, and Treatment Must Be Improved in Primary Care Clinics: There are effective approaches to monitoring and treatment that must be disseminated broadly in order to cut costs and to save lives. Dissemination efforts must focus on primary care clinics because 95% of patients with CKD have early disease and are cared for by primary care physicians (PCPs). Only 15% of patients whose estimated glomerular filtration rate (eGFR) is less than 60 mL/min/1.73m2 are aware that they have CKD, so it is especially important that PCPs become aware of the diagnosis early.5-9 Furthermore, there is evidence that CKD is under-diagnosed by PCPs. Data from our 15 primary care clinics showed that only 15% of patients with CKD had a documented diagnosis of CKD and only 40% had a urine albumin test. Hypertension Control in CKD Improves Outcomes: Hypertension (HTN) is one of the most, if not the most, important risk factor for long-term outcomes such as kidney failure, cardiovascular events, and death. A met analysis of three large cohorts of CKD patients without diabetes concluded that maintaining blood pressure below 140/90 mmHg decreases risk of these outcomes significantly.11 Several guidelines have been issued to emphasize the importance of HTN control in CKD. Evidence-based Management by PCPs for HTN in CKD: Many effective approaches for recognition of CKD and treatment of uncontrolled HTN in CKD are appropriate for the primary care setting. Lifestyle Change Counseling: Lifestyle change is recommended for all patients with uncontrolled HTN. The role of the PCP as counselor for lifestyle change is accepted and welcomed by both patients and PCPs. 15,16 Lack of time is a common barrier, but when PCPs perform brief counseling it tends to be successful, as shown in the literature on tobacco cessation. Anti-hypertensive Medication Initiation and Intensification: Evidence-based guidelines recommend certain anti-hypertensive agents in CKD, either an angiotensin converting enzyme inhibitor or angiotensin receptor blocker (ACE/ARB). The UK NICE guidelines specify a protocol for initiation and intensification of medications based on demographic characteristics.20 Efforts to simplify patients' medication regimens and provide patient education are proven to be effective in reducing blood pressure HTN in CKD Is Under-recognized and Suboptimally Managed, but CDS Has Shown Potential in Clinical Trials of the Non-CKD HTN Population: Nationally representative data show that 52% of CKD patients have diagnosed HTN, 19% have preHTN, and 16% have undiagnosed HTN. Treatment rates are suboptimal given the fact that less than 40% of CKD patients with uncontrolled HTN are prescribed anti-hypertensive medications. HTN control rates, cited as 48% to 72% across studies, are also suboptimal. A large meta-analysis of clinical decision support (CDS) for HTN in a non-CKD population showed a positive result, but with a small

average effect size of just 1 mmHg.26 An intervention in a managed care organization that incorporated CDS improved HTN control rates with an institution-wide adoption of a titration protocol and follow-up visits with a medical assistant. A multi-arm study combined CDS that recommended specific medication titration and quarterly performance reports with nurse counseling. BP control and SBP improved in all groups, but there was no significant difference between intervention groups and the control group. Another study in a non-CKD population showed a strongly positive result. The investigators tested CDS that synthesized data on the patient's current anti-hypertensive regimen and made a recommendation to intensify treatment. There was a positive result in mean BP in the arm which combined CDS with provider education and patient education (138/75 mmHg), as compared to CDS plus provider education (146/76 mmHg), and as compared to provider education alone (145/78 mmHg). Several recent trials of CDS have shown improvement in urine albumin monitoring and ACE/ARB prescription rates in CKD. However, no studies of CDS have shown an improvement in HTN management in CKD. In one pre-post study in which provider education was delivered along with multiple EHR-delivered recommendations, a flowsheet containing CKD-relevant data, and a registry, there were significant effects on diagnosis and monitoring, but no significant change in BP. 31 Another study used CDS for PCPs and nephrologists in conjunction with patient education letters and the option of a selfmanagement outreach support program. There was no impact on BP outcomes. [Sequist, personal communication] Another study compared CDS alone to CDS along with a practice improvement effort to implement the Chronic Care Model. The study found no significant effect on BP outcomes, [Fox, personal communication] The proposed study, if successful, would be the first to improve HTN in CKD patients through an intervention that incorporates CDS.

#### II. SPECIFIC AIMS

**Hypothesis:** The mean systolic blood pressure of the CKD population can be decreased by an intervention with three innovative features: 1) methods to synthesize EHR data in order to identify under-diagnosed chronic conditions, 2) iterative improvement in CDS content through human factors methods to maximize the "informativeness" of the CDS, and 3) the use of behavioral economic principles to create behavioral "nudges" internal and external to the CDS.

**Specific Aim 1:** To develop and validate the intervention.

**Specific Aim 1a:** To develop and validate the CDS that will: 1) synthesize existing laboratory tests, medication orders, and vital sign data; 2) increase recognition of CKD, 3) increase recognition of uncontrolled HTN in CKD patients; and 4) deliver evidence-based CKD and HTN management recommendations.

**Specific Aim 1b:** To improve the design and content of the CDS using human factors methods, specifically usability testing.

**Specific Aim 1c:** To develop a "wrap-around" intervention including two behavioral "nudges": 1) pre-checked default orders, and 2) an email to obtain commitment from PCPs to obtain their commitment to follow the CDS recommendations.

**Specific Aim 2:** To test the effectiveness of the intervention.

**Specific Aim 2a:** To evaluate whether the intervention developed in Aim 1 significantly decreases mean systolic blood pressure in a population of CKD patients with blood pressure > 140/90, N=2,350 (N derived from EHR data about primary care patients at 15 clinics). We will evaluate the effectiveness of the intervention in a pragmatic, cluster-randomized controlled trial, randomized at the level of the physician (185 PCPs). Secondary outcomes will include hypertension-specific process measures, such as treatment intensification.

**Specific Aim 2b:** To evaluate whether the intervention improves process measures for quality of CKD care including: documented CKD diagnosis, annual serum creatinine test, and annual urine albumin test. We will also examine process measures related to CKD care. We will use multivariable logistic regression to account for clustering by PCP using a multilevel statistical regression model, as implemented in the SAS package through the GLIMMIX procedure.

**Specific Aim 2c:** To perform a cross-over study in order to evaluate the effect of the intervention on PCP behavior and PCPs' intention to change behavior, as measured by a validated 12-item questionnaire.

#### III. SUBJECT SELECTION

**Subjects**: All patients over the age of 18 who have a visit with a PCP at one of the intervention practices during the 2 years preceding the study period will be eligible. We are able to utilize data from the past 2 years stored in the EHR to identify CKD patients with uncontrolled HTN. The first inclusion criteria will be CKD, defined as two prior eGFR 16-59 mL/min/1.73m2 separated by 90 days, as calculated by CKD-EPI, or two prior UACR >30mg/g. The second inclusion criteria will be uncontrolled hypertension, defined as at least one SBP >140 mmHg within the 2 years preceding the enrollment visit, as well as SBP >140 mmHg at the enrollment visit. Our objective was to include PCPs who have a consistent panel of primary care patients. We obtained a list of currently employed physicians, physicians assistants and nurse practitioners in our primary care network of 15 practices. We excluded residents in training, as well as physicians who were only seeing urgent care and walk-in patients.

#### **Inclusion of Women and Minorities**

Women will be represented in this study, reflecting the patient population of the BWH primary care practices and the physician population of BWH; women comprise over 50% of patients in these practices. Minorities also are fully represented in this study in proportion to their presence in these primary care practices and in proportion to their presence in the BWH physician and specialist community. The practices serve an ethnically and socioeconomically diverse patient population. Approximately 16% percent of BWH patients are Latino and 29% are Black. About 1.5% of BWH patients are Asian. Definitions of patients' race and ethnicity will be based on self-report at the time of hospital registration. By promoting uniformly high standards of patient care, our interventions may lessen disparities in care.

#### IV. SUBJECT ENROLLMENT

Randomization and Enrollment: This study will utilize a matched-pair cluster randomized design with the intervention on the cluster level, and the main outcome (6 month minus baseline change in SBP) measured at the patient level. We will have 174 clusters (made up of 185 clinicians) in the study. We will match pairs of clusters with similar number of patients and prior year mean blood pressure of patients in the cluster. One cluster in each pair with be randomized to the intervention and unit one to usual care. Patients will be electronically identified and included in the study over the course of 12 months. Patients seen by PCPs during the pilot study will be excluded. Retrospective data indicates that 70% of patients have a follow-up around 6 months. Outcomes assessment will occur at 180 days (+/- 60 days). After the 12-month enrollment period ends, data collection will continue for 6 months so that those enrolled toward the end of the enrollment period will have a full 6 months to complete any interventions ordered by the PCP. A small subset of PCPs will be enrolled in a pilot study for approximately one month, as described below in study procedures Aim 1b. Clinical outcomes will be recorded and reviewed every month over the course of the trial.

#### V. STUDY PROCEDURES

# Aim 1, and 1a Study Procedures:

Modify Rules for Automated Diagnosis of CKD and Uncontrolled HTN: Dr. Samal is a participant in the NKDEP Health Information Technology care plan working group.80 She has contributed to their efforts to new national standards for diagnosis of patients with CKD using EHR data. We will modify the rules from the MAPLE study in order to align them with this new national standard. Then, we will create rules for automated diagnosis of uncontrolled hypertension. We will implement the BPA in "silent mode" for the control arm. This means that we will identify control patients in real time according to the same inclusion criteria as intervention patients, excluding all patients who are pregnant.

Develop Rules for Evidence-based Recommendations for HTN in CKD: We will leverage past work that we have done in a study that delivered recommendations based on JNC7.73 An example of one of the rules is to determine whether anti-hypertensive agents have been prescribed but are not at highest potency. If so, the CDS will deliver a recommendation to increase the dosage. Or, if multiple agents have been prescribed at maximum potency, the CDS will access the patient's refill record. If the patient has not been refilling medications on schedule, the tool will recommend a medication adherence discussion. We will also include one-click access to documentation and orders relevant for CKD. For example, a message that gives a specific diagnosis, "This patient has stage 3b CKD with unknown level of albuminuria"), as well as an actionable order, "Click here to order a urine microalbumin to creatinine ratio test." The BPA will include a BP entry field in which a PCP can record a repeat BP reading.83,84 If the PCP enters a BP reading, it will automatically be recorded in the vital signs flowsheet and vice versa. We will include appropriate laboratory monitoring test orders. Confirmatory testing is appropriate for an abnormal urine albumin level, so we will include an order if the prior result was abnormal.85 We will also provide one-click access to print patient handouts. In order to minimize cognitive overload and improve self-efficacy we will only deliver three messages at one time. We will develop a ranked list to drive the choice of recommendations. For example, in patients with CKD and HTN who smoke, tobacco cessation would be the highest priority.

Implementation of CDS in Epic: The next step is implementation in Epic as a BPA. Each of the rules will be added to the Epic database. The BPAs appear in an area of the screen that is visible when orders are being entered. Currently, there are several cancer screening BPAs and a seasonal influenza BPA. The CDS will be moved to the Production environment in "silent mode" before the scheduled start date of the trial, where it will record when it would fire, but it will not be displayed to the user. This step will allow us to validate that the rules are accurately identifying patients and producing the correct recommendations through a chart review. We will review 10 charts of patients with CKD and uncontrolled HTN per clinic for a total of 150 charts. The CDS will be activated in the Production environment on the start date of the clinical trial in Aim 2.

<u>Validation of Hypertension-specific Process Measures</u>: In preparation for the clinical trial in Aim 2, we will validate three process measures. Two of the measures will reflect treatment intensification by the PCP, 1) an increase in dosage or 2) addition of a new anti-hypertensive agent. The third measure will reflect medication adherence by the patient using data from a pharmacy benefits manager. We will perform a retrospective chart review of 150 charts to calculate the sensitivity and specificity of each rule.

#### Aim 1b Procedure:

Task Scenario Development and Pilot Test: Usability testing clinical scenarios will be developed by two subject matter experts (Dr. Samal and Dr. Bates). Tasks will include adding CKD to the problem list, placing lab and/or medication orders, and printing patient education handouts. We will also include a test scenario that could lead the PCP to decide not to follow the CDS recommendation and we will see if they are able to enter a justification without assistance (see "accountable justification" section below). The scenarios will be reviewed by the research team to ensure that the content, format, and presentation are representative of real expected use and address the major components of the CDS. Then we will pre-load test patients with the data necessary for these scenarios and prepare the usability test procedure (described below). The usability test will be piloted with a PCP and we will ask for feedback on the usability test process, as well as content and wording of test scenarios.

<u>Usability Test Procedure:</u> A usability test plan will be developed that includes details on the testing procedure, tasks, usability metrics, usability goals, and appendices containing the test scenarios, pre-test instructions, and post-test interview questions. A moderator and observer from the research team will both attend each session. First, the moderator will describe the usability test procedure using scripted pre-test instructions to ensure that all participants receive the same instruction. The participant will be informed of the goal of evaluating the CDS and that the session will be video-taped. The moderator will describe the "think-aloud" process, asking the participant to share their thought process and expectations while completing the tasks.87 An example of think aloud will be demonstrated. Then, the moderator will begin recording the session using Morae software. The participant will read each task aloud, attempt the task, and inform the moderator when the task is complete. The moderator will record task success or failure based on the intended outcome as described in the test plan. If a participant is having trouble completing a task, he or she will be given an assist at the moderator's discretion. The observer will make note of assists and other usability or comprehension issues that arise. After all tasks are complete, the moderator will administer a verbal post-test interview. The moderator will ask questions like, "How did you interpret this?", "Why did

you do X?" and "What would you change about the content of the CDS?" The moderator and observer will manually record observations during the testing session. In addition to the comments and data recorded during the session, usability metrics will be coded after the session using Morae software. Usability metrics are measurements collected to determine to what extent usability goals have been met. The metrics will include task completion success rates, time-on-task, error rates, and assists by the moderator. We will be able to compare these measurements to those gathered from subsequent tests to determine whether iterative changes to the CDS have improved the usability of the CDS. Qualitative analysis: Qualitative methods will be employed to analyze the data. The research assistant will review the video recordings to identify usability issues based on observations of the participants during the task and the participants' think-aloud comments. Video recordings will be transcribed verbatim, and subject identifiers will be removed from the transcripts. The transcripts will be organized by task and participant and then quotes will be identified that illustrate a user expectation, frustration, or misinterpretation of content or functionality.

<u>Pilot Study</u>: Prior to the clinical trial, a pilot study will be conducted in live clinical settings. A subgroup of PCPs will be selected an the BPAs will be turned on for approximately one month. Interaction with the BPAs will be monitored. Each time a BPA fires the research team will contact the PCP by email to gather feedback through surveys and/or interviews. Iterative refinement of BPAs may be undertaken.

#### Aim 1c Procedure:

- 1) Pre-checked, no-action default: The first nudge will be part of the CDS. We will display the CDS with certain options pre-selected. We plan to include addition of the CKD diagnosis to the problem list and addition of a patient education handout to the after-visit summary.
- 2) Pledge email to obtain commitment from PCPs to follow the CDS recommendations: As a starting point, we need to ensure that PCPs are aware of the clinical practice guidelines. At the beginning of the study, we will send an advertisement email to all PCPs in the network. In addition, as part of the intervention, we will ask PCPs to commit to following the recommendations presented to them in the BPA, or writing their rationale in the CDS if they choose not to. The PI will send an email via REDCap to intervention PCPs giving a brief overview of the CDS content. By clicking a link in the email, the intervention PCP will come to a REDCap survey asking them to type their name to pledge to consider the CDS recommendations provided in our BPAs. The control PCPs will receive a similar email without the specific details about our study and without the REDCap link.

Behavioral Science Methods Review Committee: Though the research team does include co-investigators with expertise in behavioral science methods, we have decided to convene an advisory group consisting of three experts in behavioral science as applied in interventions for both PCPs and patients. We have chosen the members of this committee based upon their familiarity with chronic disease management interventions and EHR-based interventions. We have limited the group to three members because we plan to meet on a monthly basis during the first two years of the study. This group will give advice to the research team on elements of Aim 1 and the roll-out of the clinical trial.

#### **Specific Aim 2 & 2a Procedures:**

<u>Setting</u>: The Brigham and Women's Primary Care Practice-Based Research Network (BWPC PBRN) is one of 155 PBRNs nationally certified by the Agency for Healthcare Research and Quality (AHRQ). The BWPC PBRN is a network of 15 practices which includes hospital-based practices, community-based practices, and community health centers affiliated with Brigham and Women's Hospital. The network includes 185 primary care physicians that care for approximately 150,000 patients.

<u>Subjects</u>: All patients over the age of 18 who have a visit with a PCP at one of the intervention practices during the 2 years preceding the study period will be eligible. We are able to utilize data from the past five years stored in the EHR to identify CKD patients with uncontrolled HTN. The first inclusion criteria will be CKD, defined as two prior eGFR 16-59 mL/min/1.73m<sub>2</sub> separated by 90 days, as calculated by CKD-EPI, or two prior UACR >30mg/g. The second inclusion criteria will be uncontrolled hypertension, defined as at least two SBP >140 mmHg within the 2 years preceding the study period. We will exclude all patients who are currently pregnant. The CDS will review lab data starting five years before the visit to determine whether the patient has CKD using the logic described above. If the patient has CKD, the CDS will search BP data starting one year before the visit to determine whether the patient has had at least two SBP > 140 mmHg.

#### Specific Aim 2b Procedure:

<u>Outcomes</u>: We will analyze the actual use of the CDS, defined as interaction with the BPA, signing of orders, or accountable justification documentation within the BPA.

#### VI. BIOSTATISTICAL ANALYSIS

Data collected during the pilot study will not be included in the final analysis. Patients enrolled in the pilot study will not be enrolled in the final analysis. However, PCPs in the pilot study will be included in the intervention arm of the main clinical trial. A subgroup analysis will be performed on patients of these PCPs.

Table 1. Outcome Variables and Measures for Both Arms

| Measurement<br>Variable | Form of Variable | Analysis Metric | Time Point |
|---|---|---|---|
| Primary | | | |
| Mean SBP | Continuous | Change from baseline | 6 months, 12 months, 18 months |
| Secondary | | | |
| Controlled SBP<br>Rate | Dichotomous | Proportion of patients with controlled SBP rate | 6 months, 12 months, 18 months |
| Urine Albumin to<br>Creatinine Ratio | Continuous | Urine Albumin to Creatinine Ratio | 6 months, 12<br>months, 18 months |
| Serum Creatinine > 2.0 | Dichotomous | Proportion of patients with Creatinine > 2.0 | Monthly |
| eGFR | Continuous | eGFR | 6 months, 12 months, 18 months |

| Medication ordered | Dichotomous | Proportion of patients with recommended medication ordered | 6 months |
|---|---|---|---|
| Basic metabolic panel ordered | Dichotomous | Proportion of patients with basic metabolic panel ordered | 6 months |
| Referral to e-<br>consults | Dichotomous | Proportion of patients with referral to e-consults | 6 months |
| BPA acceptance | Dichotomous | Proportion of patients where BPA was accepted | 6 months |
| Mean SBP of less<br>than 110 | Dichotomous | Proportion of patients with mean SBP of less than 110 | Monthly |
| Newly documented allergy | Dichotomous | Proportion of patients with newly documented allergy due to adverse drug events | Monthly |
| K+ > 5.2 | Dichotomous | Proportion of patients with K+ > 5.2 | Monthly |
| K+ < 3.6 | Dichotomous | Proportion of patients with K+ < 3.6 | Monthly |
| Mean SBP intent-<br>to-intervene<br>analysis with<br>imputation of<br>missing 6-month BP<br>measurement | Dichotomous | Proportion of patients with missing 6-month BP measurement | 6 months |
| Controlled SBP Rate intent-to- intervene analysis with imputation of missing 6-month BP measurement | Dichotomous | Proportion of patients with missing 6-month BP measurement | 6 months |

Table 2. Outcome Variables and Measures for Intervention Arm Only

| Measurement | Form of Variable | Analysis Metric | Time Point |
|---|---|---|---|
| Variable Acknowledgment reason entered | Dichotomous | Proportion of patients with acknowledgment reason entered | 6 months |
| Feedback button clicked | Dichotomous | Proportion of patients with feedback button clicked | 6 months |
| PCP participation on pledge email survey | Dichotomous | Proportion of patients whose PCPs participated in pledge email survey | 6 months |
| Guideline accessed | Dichotomous | Proportion of patients with guideline accessed | 6 months |

# VII. RISKS AND DISCOMFORTS

There are minimal risks to physicians or patients as a result of the intervention. For clinicians, there is a risk that the decision support and other tools could have unexpected adverse consequences such as creation of more work, unfavorable workflow issues, and overdependence on technology. Although important to consider, these risks are balanced by evidence suggesting the effectiveness of computerized clinical decision support to improve the quality of patient care. For patients, the risks are those that are typically undertaken in the receipt of general medical care. That is, it is conceivable that the intervention could result in a change in management (e.g., ordering more tests, referral), but in the case of chronic kidney disease this may in fact lead to a clinical benefit. There also is the possibility of psychological risk to patients associated with being labeled as having chronic kidney disease; however, this risk is outweighed by the potential benefits associated with better evaluation and treatment of the disease. Finally, there is a risk of overtreatment of hypertension which may cause hypotension or an acute decrease in kidney function. The intervention is delivered to the primary care physician, who will weigh the risk and benefit of treatment intensification. However, this risk is expected to be low since we only recommend treatment intensification within consensus guidelines.

#### VIII. POTENTIAL BENEFITS

This research has the potential benefit of improving the quality of care for patients in the intervention practices, which ultimately could prevent disease progression and death. There are no potential benefits to the control subjects, who will receive current standard of care.

# IX. MONITORING AND QUALITY ASSURANCE

The investigators will establish an independent Data Safety Monitoring Board (DSMB), which will serve as an independent group to monitor participant safety, study burden and scientific validity of the clinical data. The PI will ensure that the research is conducted in an ethical manner in accordance with good clinical practice and meets all applicable regulatory laws and policies. In addition to meeting the responsibilities for protecting the rights, safety, and welfare of the subjects enrolled in the research, the PI will review safety data, study conduct, procedural safety enrollment, adverse events, and other study-related information. The PI and co-investigators will review enrollment, adverse events and any recent literature that may be relevant to the research on a quarterly basis. Formal minutes with discussion points and remediation/actions plans (e.g. changes to protocol and consent documents) will be created, maintained, and relayed to the DSMB. The DSMB will convene in person or by teleconference once per year. At this meeting, the board will review any cases where systolic blood pressure was found to be below 110 mmHg, any reported adverse events, and deaths of enrolled patients.

# X. REFERENCES

1. Coresh J, Selvin E, Stevens LA, et al. Prevalence of chronic kidney disease in the United States. *JAMA*. 2007;298(17):2038-2047.

- 2. Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. *N Engl J Med*. 2004;351(13):1296-1305.
- 3. Hirth RA. The organization and financing of kidney dialysis and transplant care in the United States of America. *Int J Health Care Finance Econ.* 2007;7(4):301-318.
- 4. USRDS 2009 Annual Data Report: Atlas of End-Stage Renal Disease in the United States. National Institutes of Health, Bethesda, MD;2009.
- 5. Plantinga LC, Tuot DS, Powe NR. Awareness of chronic kidney disease among patients and providers. *Adv Chronic Kidney Dis May.* 2010;17(3):225-236.
- 6. USRDS 2011 Annual Data Report: Atlas of End-Stage Renal Disease in the United States. National Institutes of Health, Bethesda, MD;2011.
- 7. Tuot DS, Powe NR. Chronic Kidney Disease in Primary Care: An Opportunity for Generalists. *Journal of general internal medicine*. 2011.
- 8. Parker MG, Ibrahim T, Shaffer R, Rosner MH, Molitoris BA. The Future Nephrology Workforce: Will There Be One? *Clinical journal of the American Society of Nephrology : CJASN.* 2011.
- 9. Pellegrino B, Schmidt RJ. Why Work Together? Developing Effective Comanagement Strategies for the Care of Patients With CKD. *Advances in chronic kidney disease*. 2011;18(6):396-399.
- 10. Samal L, Linder JA, Bates DW, Wright A. Electronic problem list documentation of chronic kidney disease and quality of care. *BMC Nephrol*. 2014;15:70.
- 11. Upadhyay A, Earley A, Haynes SM, Uhlig K. Systematic review: blood pressure target in chronic kidney disease and proteinuria as an effect modifier. *Ann Intern Med.* 2011;154(8):541-548.
- 12. Kidney Disease: Improving Global Outcomes CKDWG. KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. *Kidney Int. Suppl.* 2013;3(Journal Article):1-150.
- 13. James PA, Oparil S, Carter BL, et al. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). *JAMA*. 2014;311(5):507-520.
- 14. Taler SJ, Agarwal R, Bakris GL, et al. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for management of blood pressure in CKD. *Am J Kidney Dis*. 2013;62(2):201-213.

- 15. Wechsler H, Levine S, Idelson RK, Schor EL, Coakley E. The physician's role in health promotion revisited--a survey of primary care practitioners. *N Engl J Med*. 1996;334(15):996-998.
- 16. Levine DM. The physician's role in health-promotion and disease prevention. *Bull N Y Acad Med.* 1987;63(10):950-956.
- 17. Ashenden R, Silagy C, Weller D. A systematic review of the effectiveness of promoting lifestyle change in general practice. *Fam Pract.* 1997;14(2):160-176.
- 18. Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. *JAMA*. 1988;259(19):2883-2889.
- 19. Mullen PD, Simons-Morton DG, Ramirez G, Frankowski RF, Green LW, Mains DA. A meta-analysis of trials evaluating patient education and counseling for three groups of preventive health behaviors. *Patient Educ Couns.* 1997;32(3):157-173.
- 20. McCormack T, Krause T, O'Flynn N. Management of hypertension in adults in primary care: NICE guideline. *Br J Gen Pract*. 2012;62(596):163-164.
- 21. Glynn LG, Murphy AW, Smith SM, Schroeder K, Fahey T. Interventions used to improve control of blood pressure in patients with hypertension. *Cochrane Database Syst Rev.* 2010(3):CD005182.
- 22. Crews DC, Plantinga LC, Miller ER, 3rd, et al. Prevalence of chronic kidney disease in persons with undiagnosed or prehypertension in the United States. *Hypertension*. 2010;55(5):1102-1109.
- 23. Sonawane KB, Qian J, Hansen RA. Utilization patterns of antihypertensive drugs among the chronic kidney disease population in the United States: a cross-sectional analysis of the national health and nutrition examination survey. *Clin Ther*. 2015;37(1):188-196.
- 24. Plantinga LC, Miller ER, 3rd, Stevens LA, et al. Blood pressure control among persons without and with chronic kidney disease: US trends and risk factors 1999-2006. *Hypertension*. 2009;54(1):47-56.
- 25. Muntner P, Anderson A, Charleston J, et al. Hypertension awareness, treatment, and control in adults
- with CKD: results from the Chronic Renal Insufficiency Cohort (CRIC) Study. *Am J Kidney Dis*.

2010;55(3):441-451.

- 26. Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. *Cochrane Database Syst Rev.* 2009;(3)(3):CD001096.
- 27. Jaffe MG, Lee GA, Young JD, Sidney S, Go AS. Improved blood pressure control associated with a large-scale hypertension program. *JAMA*. 2013;310(7):699-705.
- 28. Bosworth HB, Olsen MK, Dudley T, et al. Patient education and provider decision support to control blood pressure in primary care: a cluster randomized trial. *Am Heart J.* 2009;157(3):450-456.
- 29. Roumie CL, Elasy TA, Greevy R, et al. Improving blood pressure control through provider education, provider alerts, and patient education: a cluster randomized trial. *Ann Intern Med.* 2006;145(3):165-175.
- 30. Abdel-Kader K, Fischer GS, Li J, Moore CG, Hess R, Unruh ML. Automated clinical reminders for primary care providers in the care of CKD: a small cluster-randomized controlled trial. *Am J Kidney Dis.* 2011;58(6):894-902.
- 31. Litvin CB, Hyer JM, Ornstein SM. Use of Clinical Decision Support to Improve Primary Care Identification and Management of Chronic Kidney Disease (CKD). *J Am Board Fam Med.* 2016;29(5):604-612.
- 32. Fox CH, Vest BM, Kahn LS, et al. Improving evidence-based primary care for chronic kidney disease: study protocol for a cluster randomized control trial for translating evidence into practice (TRANSLATE CKD). *Implement Sci.* 2013;8(88).
- 33. Cabana MD, Rand CS, Powe NR, et al. Why don't physicians follow clinical practice guidelines? A framework for improvement. *JAMA*. 1999;282(15):1458-1465
- 34. Lea JP, McClellan WM, Melcher C, Gladstone E, Hostetter T. CKD risk factors reported by primary care physicians: do guidelines make a difference? *Am J Kidney Dis.* 2006;47(1):72-77.
- 35. Ostbye T, Yarnall KS, Krause KM, Pollak KI, Gradison M, Michener JL. Is there time for management of patients with chronic diseases in primary care? *Ann Fam Med.* 2005;3(3):209-214.
- 36. Bolen SD, Bricker E, Samuels TA, et al. Factors associated with intensification of oral diabetes medications in primary care provider-patient dyads: a cohort study. *Diabetes Care.* 2009;32(1):25-31.
- 37. Parchman ML, Pugh JA, Romero RL, Bowers KW. Competing demands or clinical inertia: the case of elevated glycosylated hemoglobin. *Ann Fam Med.* 2007;5(3):196-201. 38. Rocco MV, Cheung AK. A SPRINT to the finish, or just the beginning? Implications of the SPRINT results for nephrologists. *Kidney Int.* 2016;89(2):261-263.

- 39. Allen AS, Forman JP, Orav EJ, Bates DW, Denker BM, Sequist TD. Primary care management of chronic kidney disease. *J Gen Intern Med.* 2011;26(4):386-392.
- 40. Fox CH, Swanson A, Kahn LS, Glaser K, Murray BM. Improving chronic kidney disease care in primary care practices: an upstate New York practice-based research network (UNYNET) study. *J Am Board Fam Med.* 2008;21(6):522-530.
- 41. Samal L, D'Amore JD, Bates DW, Wright A. Implementation of a Scalable, Webbased, Automated Clinical Decision Support Risk Prediction Tool for Chronic Kidney Disease Using C-CDA and Application Programming Interfaces. *J Am Med Inform Assoc.* 2017;[in press].
- 42. Tangri N, Grams ME, Levey AS, et al. Multinational Assessment of Accuracy of Equations for Predicting Risk of Kidney Failure: A Meta-analysis. *JAMA*. 2016;315(2):164-174.
- 43. Tangri N, Stevens LA, Griffith J, et al. A predictive model for progression of chronic kidney disease to kidney failure. *JAMA*. 2011;305(15):1553-1559.
- 44. Feblowitz JC, Wright A, Singh H, Samal L, Sittig DF. Summarization of clinical information: a conceptual model. *J Biomed Inform*. 2011;44(4):688-699.
- 45. Schnipper JL, Linder JA, Palchuk MB, Einbinder JS LQ, Postilnik A, Middleton B. "Smart forms" in an electronic medical record: Documentation-based clinical decision support to improve disease management. *J Am Med Inform Assoc.* 2008;15(4):513-523.
- 46. Hicks LS, Malley AJ, Lieu TA, Keegan T. MBJ, Guadagnoli E., Landon B.E. Impact of health disparities collaboratives on racial/ethnic and insurance disparities in US community health centers. *Arch Intern Med.* 2010;170(3):279-286.
- 47. Murray MD, Harris LE, Overhage JM, et al. Failure of computerized treatment suggestions to improve health outcomes of outpatients with uncomplicated hypertension: results of a randomized controlled trial. *Pharmacotherapy*. 2004;24(3):324-337.
- 48. Linder JA, Rigotti NA, Schneider LI, et al. Clinician characteristics and use of novel electronic health record functionality in primary care. *J Am Med Inform Assoc.* 2011;18 Suppl 1:i87-90.
- 49. Sittig DF, Krall MA, Dykstra RH, Russell A, Chin HL. A survey of factors affecting clinician acceptance of clinical decision support. *BMC Med Inform Decis Mak*. 2006;6(6).
- 50. Karsh BT, Weinger MB, Abbott PA, Wears RL. Health information technology: fallacies and sober realities. *J Am Med Inform Assoc.* 2010;17(6):617-623.

- 51. Kushniruk AW, Patel VL. Cognitive and usability engineering methods for the evaluation of clinical information systems. *J Biomed Inform*. 2004;37(1):56-76.
- 52. Rayo MF, Moffatt-Bruce SD. Alarm system management: evidence-based guidance encouraging direct measurement of informativeness to improve alarm response. *BMJ Qual Saf.* 2015;24(4):282-286.
- 53. Lees MN, Lee JD. The influence of distraction and driving context on driver response to imperfect collision warning systems. *Ergonomics*. 2007;50(8):1264-1286.
- 54. Gosbee JW. Conclusion: You need human factors engineering expertise to see design hazards that are hiding in "plain sight!". *Jt Comm J Qual Saf.* 2004;30(12):696-700.
- 55. Ash JS, Sittig DF, Poon EG, Guappone K, Campbell E, Dykstra RH. The extent and importance of unintended consequences related to computerized provider order entry. *J Am Med Inform Assoc.* 2007;14(4):415-423.
- 56. Bates DW, Kuperman GJ, Wang S, et al. Ten commandments for effective clinical decision support: making the practice of evidence-based medicine a reality. *J Am Med Inform Assoc.* 2003;10(6):523-530.
- 57. Ariely D. *Predictably irrational: The hidden forces that shape our decisions*. New York: Harper Perennial; 2010.
- 58. Johnson EJ, Goldstein D. Medicine. Do defaults save lives? *Science*. 2003;302(5649):1338-1339.
- 59. Halpern SD, Loewenstein G, Volpp KG, et al. Default options in advance directives influence how patients set goals for end-of-life care. *Health Aff (Millwood)*. 2013;32(2):408-417.
- 60. Malhotra S, Ancker JS, Gossey JT, Cole CL, Kaushal R, Cheriff AD. Promoting generic medication prescribing by order interface redesign: small change, large impact. *Stud Health Technol Inform.* 2012;180:1194-1196.
- 61. Malhotra S, Cheriff AD, Gossey JT, Cole CL, Kaushal R, Ancker JS. Effects of an e-Prescribing interface redesign on rates of generic drug prescribing: exploiting default options. *J Am Med Inform Assoc.* 2016;23(5):891-898.
- 62. Loewenstein GB, C; Hagmann, D. Warning: You Are About to Be Nudged. *Behavioral Science & Policy*. 2014;1(1):35-42.
- 63. Meeker D, Knight TK, Friedberg MW, et al. Nudging guideline-concordant antibiotic prescribing: a randomized clinical trial. *JAMA Intern Med.* 2014;174(3):425-431.

- 64. Meeker D, Linder JA, Fox CR, et al. Effect of Behavioral Interventions on Inappropriate Antibiotic Prescribing Among Primary Care Practices: A Randomized Clinical Trial. *JAMA*. 2016;315(6):562-570.
- 65. Lerner JS, Tetlock PE. Accounting for the effects of accountability. *Psychol Bull*. 1999;125(2):255-275.
- 66. Milinski M, Semmann D, Krambeck HJ. Reputation helps solve the 'tragedy of the commons'. *Nature*. 2002;415(6870):424-426.
- 67. Cialdini R, Reno R, Kallgren C. A focus theory of normative conduct: recycling the concept of norms to reduce littering in public places. *J Pers Soc Psychol*. 1990;58(5):1015-1026.
- 68. De Cremer D, Barker M. Accountability and cooperation in social dilemmas: the influence of others' reputational concerns. *Curr Psychol.* 2003;22(2):155-163.
- 69. Persell SD, Doctor JN, Friedberg MW, et al. Behavioral interventions to reduce inappropriate antibiotic prescribing: a randomized pilot trial. *BMC Infect Dis.* 2016;16:373.
- 70. Samal L, Wright A, Waikar SS, Linder JA. Nephrology co-management versus primary care solo management for early chronic kidney disease: a retrospective cross-sectional analysis. *BMC Nephrol*. 2015;16:162.
- 71. Wright A, Pang J, Feblowitz JC, et al. Improving completeness of electronic problem lists through clinical decision support: A randomized, controlled trial. *J Am Med Inform Assoc.* 2012;19(4):555-561.
- 72. Linder JA, Schnipper JL, Tsurikova R, et al. Electronic health record feedback to improve antibiotic prescribing for acute respiratory infections. *Am J Manag Care*. 2010;16(12 Suppl HIT):e311-319.
- 73. Hicks LS, Sequist TD, Ayanian JZ, et al. Impact of computerized decision support on blood pressure management and control: a randomized controlled trial. *J Gen Intern Med*. 2008;23(4):429-441.
- 74. Sequist TD, Gandhi TK, Karson AS, et al. A randomized trial of electronic clinical reminders to improve quality of care for diabetes and coronary artery disease. *J Am Med Inform Assoc.* 2005;12(4):431-437.
- 75. Linder JA, Rigotti NA, Schneider LI, Kelley JH, Brawarsky P, Haas JS. An electronic health recordbased intervention to improve tobacco treatment in primary care: a cluster-randomized controlled trial. *Arch Intern Med.* 2009;169(8):781-787.

- 76. Hsu CY, Bates DW, Kuperman GJ, Curhan GC. Diabetes, hemoglobin A(1c), cholesterol, and the risk of moderate chronic renal insufficiency in an ambulatory population. *Am J Kidney Dis.* 2000;36(2):272-281.
- 77. Hsu CY, Bates DW, Kuperman GJ, Curhan GC. Blood pressure and angiotensin converting enzyme inhibitor use in hypertensive patients with chronic renal insufficiency. *Am J Hypertens*. 2001;14(12):1219-1225.
- 78. Hsu CY, Bates DW, Kuperman GJ, Curhan GC. Relationship between hematocrit and renal function in men and women. *Kidney Int.* 2001;59(2):725-731.
- 79. Chertow GM, Lee J, Kuperman GJ, et al. Guided medication dosing for inpatients with renal insufficiency. *JAMA*. 2001;286(22):2839-2844.
- 80. NKDEP Health Information Technology Working Group. 2017; https://www.niddk.nih.gov/healthinformation/health-communication-programs/nkdep/working-groups/health-information-technologyworking-group/Pages/default.aspx. Accessed May 30, 2017.
- 81. Drawz PE, Archdeacon P, McDonald CJ, et al. CKD as a Model for Improving Chronic Disease Care through Electronic Health Records. *Clin J Am Soc Nephrol*. 2015;10(8):1488-1499.
- 82. Matsushita K, Selvin E, Bash LD, Astor BC, Coresh J. Risk implications of the new CKD Epidemiology Collaboration (CKD-EPI) equation compared with the MDRD Study equation for estimated GFR: the Atherosclerosis Risk in Communities (ARIC) Study. *Am J Kidney Dis.* 2010;55(4):648-659.
- 83. Meeker D, Linder JA, Fox CR, Friedberg MW, Persell, S.D., Goldstein, N.J., Knight, T.K., Hay, J.W., Doctor, J.N. Effect of behavioral interventions on inappropriate antibiotic prescribing among primary care practices: A randomized clinical trial. *JAMA*. 2016;315(6):562-570.
- 84. Persell SD, Dolan NC, Friesema EM, Thompson JA, Kaiser D, Baker DW. Frequency of inappropriate medical exceptions to quality measures. *Ann Intern Med*. 2010;152(4):225-231.
- 85. KDIGO clinical practice guideline for the evaluation and management of chronic kidney disease. *Kidney Int Suppl 1*. 2013;3(1).
- 86. Regalado M, Yang S, Wesson DE. Cigarette smoking is associated with augmented progression of renal insufficiency in severe essential hypertension. *Am J Kidney Dis.* 2000;35(4):687-694.
- 87. Jaspers MW, Steen T, van den Bos C, Geenen M. The think aloud method: a guide to user interface design. *Int J Med Inform.* 2004;73(11-12):781-795.

- 88. Singh K, Waikar SS, Samal L. Evaluating the feasibility of the KDIGO CKD referral recommendations. *BMC Nephrol*. 2017;18(1):223.
- 89. Natarajan S, Lipsitz SR, Fitzmaurice GM, et al. An extension of the Wilcoxon Rank-Sum test for complex sample survey data. *J R Stat Soc Ser C Appl Stat.* 2012;61(4):653-664.
- 90. Legare F, Borduas F, Jacques A, et al. Developing a theory-based instrument to assess the impact of continuing professional development activities on clinical practice: a study protocol. *Implement Sci.* 2011;6:17.
- 91. Legare F, Borduas F, Freitas A, et al. Development of a simple 12-item theory-based instrument to assess the impact of continuing professional development on clinical behavioral intentions. *PLoS One.* 2014;9(3):e91013.
- 92. Legare F, Freitas A, Turcotte S, et al. Responsiveness of a simple tool for assessing change in behavioral intention after continuing professional development activities. *PLoS One.* 2017;12(5):e0176678.